CLINICAL TRIAL: NCT02840578
Title: Measurement of NK Cell Activity in Whole Blood in Subjects Being Screened for Lung Cancer
Brief Title: NK Cell Activity in Smokers Screened for Lung Cancer
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: ATGen Global (Unknown)
Responsible Party: Principal Investigator, Christopher Lee, Associate Professor, University of Southern California
Other Study IDs: NK Cell Activity
Record Dates: First submitted 2016-07-14; First posted 2016-07-21 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample (1 ml) will be collected following a set of established Standard Operating Procedures (SOPs). Blood samples will be incubated for 20 hours after initial draw then centrifuged. Serum will then be frozen and stored at USC until they are sent to Cynvenio's CLIA and CAP certified laboratory in Thousand Oaks, CA for ELISA processing. All serum samples will be picked up by a Cynvenio representative who will personally deliver the specimens to the Cynvenio Labs.
Oversight: Data Monitoring Committee: No

SUMMARY:
Objectives: To examine whether NK cell activity associates with two confirmed risk factors: (1) presence of indeterminate lung nodule(s) and (2) smoking exposure after controlling for potential confounders, including age, gender, body mass index (BMI), personal history of any cancer, and family history of cancer. This project is aimed at measuring NK cell activity, which may eventually help in reducing false positive rates of LDCT screening, improve early detection of lung cancer, and assist in risk assessment in patients with lung cancer. The investigators hypothesize that measurement of NK cell activity may be a useful tool for assessing changes in immunosurveillance in patients with conditions or diseases where NK cell activity has been shown to be reduced, such as lung cancer

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer mortality in the United States. Despite considerable clinical research in multi-modality cancer treatment, there has been no significant decrease in lung cancer-specific mortality over the past three decades. The recent results of the National Lung Screening Trial (NLST) established that screening high-risk individuals using low-dose CT (LDCT) significantly reduces lung cancer-related mortality. One caveat is that approximately 96% of the "positive" results in the NLST were found not to be related to lung cancer. The difficulty in determining which subjects with suspicious lesions should be biopsied or operated on could be alleviated by the development of highly specific lung cancer biomarkers that could complement LDCT. Thus, novel, complementary, non-invasive diagnostic tools with high sensitivity and specificity would clearly be of enormous benefit to patients with a "positive" screening exam. This study will look at measuring the activity of natural killer (NK) cells using the in vitro diagnostic device NK Vue™ in a cohort of current and former smokers (n=100) who meet the criteria for LDCT screening established by the National Comprehensive Cancer Network (NCCN) as a result of the positive findings from the NLST. This project is aimed at measuring the NK cell activity, which may eventually help in reducing false positive rates of LDCT screening, improve early detection of lung cancer, and assist in risk assessment in patients with lung cancer. The Investigators hypothesize that measurement of NK cell activity may be a useful tool for assessing changes in immunosurveillance in patients with conditions or diseases where NK cell activity has been shown to be reduced, such as lung cancer.

Objectives Specific Aim 1: To examine whether NK cell activity associates with two confirmed risk factors: (1) presence of indeterminate lung nodule(s) and (2) smoking exposure after controlling for potential confounders, including age, gender, body mass index (BMI), personal history of any cancer, and family history of cancer.

Specific Aim 2 (Exploratory): In the study cohort, investigators expect approximately 45% of patients having at least one indeterminate lung nodule. Among those with lung nodule(s), investigators will examine whether NK cell activity associates with size of the largest lung nodule after controlling for potential confounders, including smoking exposure, age, gender, BMI, personal history of any cancer, and family history of cancer

ELIGIBILITY:
Inclusion Criteria:

* At the time of registration, subjects must have a current or previous cumulative cigarette smoking history of ≥ 20 pack years (packs per day multiplied by the number of years smoked). If smoking history is between 20 and 29 pack years, subjects must have an additional risk factor (i.e. radon exposure, occupational exposure, personal history of smoking-associated cancer, family history of lung cancer in first-degree relatives, COPD or pulmonary fibrosis).
* At the time of registration former smokers without additional risk factor(s) must have quit smoking within the preceding 15 years.
* Subjects must be willing to provide blood samples as biospecimens for the study.
* At the time of registration, subjects must have recovered from the toxic effects of prior therapy: ≥6 months (182 days) from the last dose of prior cytotoxic therapy.
* At the time of registration, subjects must have recovered from the effects of prior pneumonia or acute respiratory infection treated by antibiotics by a physician: ≥12 weeks (84 days) from the first dose of antibiotics.

Exclusion Criteria:

* Medical or psychiatric condition precluding informed medical consent.
* Prior history of lung cancer.
* Treatment for or advisement by a physician of evidence of any cancer within the past five years, with the exceptions of non-melanoma skin cancer and most in-situ carcinomas. (Treatment for, or evidence of, melanoma or in-situ bladder/transition cell carcinomas within the preceding five years renders the potential participant ineligible.)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects must be ages 50 to 80 years and 364 days, and are males or females not of childbearing potential.
Sampling Method: Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
The association between NK cell activity and presence of lung nodule and smoking exposure (pack-years), | 1 year
  Multivariate generalized linear model will be used to examine the association controlling for potential confounders including age, gender, BMI, personal history of any cancer, and family history of cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Lee, MD, Principal Investigator — University of Southern California
Locations (1):
- USC Department of Radiology, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] Lee SB, Cha J, Kim IK, Yoon JC, Lee HJ, Park SW, Cho S, Youn DY, Lee H, Lee CH, Lee JM, Lee KY, Kim J. A high-throughput assay of NK cell activity in whole blood and its clinical application. Biochem Biophys Res Commun. 2014 Mar 14;445(3):584-90. doi: 10.1016/j.bbrc.2014.02.040. Epub 2014 Feb 18. PMID 24561245
- [Background] Koo KC, Shim DH, Yang CM, Lee SB, Kim SM, Shin TY, Kim KH, Yoon HG, Rha KH, Lee JM, Hong SJ. Reduction of the CD16(-)CD56bright NK cell subset precedes NK cell dysfunction in prostate cancer. PLoS One. 2013 Nov 4;8(11):e78049. doi: 10.1371/journal.pone.0078049. eCollection 2013. PMID 24223759